CLINICAL TRIAL: NCT05595369
Title: RECOVER-VITAL: A Platform Protocol for Evaluation of Interventions for Viral Persistence, Viral Reactivation, and Immune Dysregulation in Post-Acute Sequelae of SARS-CoV-2 Infection (PASC)
Brief Title: RECOVER-VITAL: Platform Protocol to Measure the Effects of Antiviral Therapies on Long COVID Symptoms
Acronym: RECOVER-VITAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kanecia Obie Zimmerman (Other)
Responsible Party: Sponsor-Investigator, Kanecia Obie Zimmerman, Associate Professor of Pediatrics, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00111697; OTA-21-015G (Other Grant/Funding Number: NIH grant to RTI; RTI subcontracting with DCRI)
Record Dates: First submitted 2022-10-11; First posted 2022-10-27 (Actual); Results first posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Long COVID; Long Covid19
Keywords: PASC
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Intervention Model Description: As part of screening, potential participants will answer symptom questions. Eligible participants will then complete relevant Symptom Cluster assessments at the Screening visit. Participants will subsequently be assigned to one of the three Symptom Clusters based on the assessments. Participants must meet certain criteria within a specific symptom cluster in order to be included in the cluster. After study enrollment and initial cluster assignment, further assessments will be performed. Participants will undergo assessments for the symptom clusters for which the participants qualify.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Experimental: Paxlovid 25 day dosing (Experimental): Drug: Paxlovid 25 day dosing Paxlovid (nirmatrelvir 300mg, ritonavir 100mg) bid x 25 days See NCT05965726 (Paxlovid Sub-study)
  Interventions: Drug: Experimental: Paxlovid 25 day dosing
- Experimental: Paxlovid 15 day dosing (Experimental): Drug: Paxlovid 15 day Dosing Paxlovid (nirmatrelvir 300mg and ritonavir 100mg) bid x 15 days then ritonavir 100mg bid plus nirmatrelvir matching placebo bid x 10 days See NCT05965726 (Paxlovid Sub-study)
  Interventions: Drug: Experimental: Paxlovid 15 day dosing
- Placebo Comparator: Control (Placebo Comparator): Drug: Control ritonavir 100mg taken bid plus nirmatrelvir matching placebo bid bid x 25 days See NCT05965726 (Paxlovid Sub-study)
  Interventions: Drug: Placebo Comparator: Control

INTERVENTIONS:
Drug: Experimental: Paxlovid 25 day dosing — Drug: Paxlovid 25 day dosing Paxlovid (nirmatrelvir 300mg, ritonavir 100mg) bid x 25 days See NCT05965726 (Paxlovid Sub-study)
  Arms: Experimental: Paxlovid 25 day dosing
Drug: Experimental: Paxlovid 15 day dosing — Drug: Paxlovid 15 day Dosing Paxlovid (nirmatrelvir 300mg and ritonavir 100mg) bid x 15 days then ritonavir 100mg bid plus nirmatrelvir matching placebo bid x 10 days See NCT05965726 (Paxlovid Sub-study)
  Arms: Experimental: Paxlovid 15 day dosing
Drug: Placebo Comparator: Control — Drug: Control ritonavir 100mg taken bid plus nirmatrelvir matching placebo bid bid x 25 days See NCT05965726 (Paxlovid Sub-study)
  Arms: Placebo Comparator: Control

SUMMARY:
This study is a platform protocol designed to be flexible so that it is suitable for a wide range of settings within health care systems and in community settings where it can be integrated into COVID-19 programs and subsequent treatment plans. This protocol is a prospective, multi-center, multi-arm, double-blind, randomized, controlled platform trial with different interventions organized as appendices to the protocol. Each appendix (or sub-study) evaluates potential mechanisms of action, efficacy, and safety of antivirals and other therapeutics in individuals with PASC, according to the platform protocol objectives. The hypothesis is that persistent viral infection, viral reactivation, and/or overactive/chronic immune response and inflammation are underlying contributors to PASC and that antiviral and other applicable therapies may result in viral clearance or decreased inflammation and improvement in PASC symptoms.

DETAILED DESCRIPTION:
Participants will be randomized to study interventions or placebo/controls based on the arms that are actively enrolling at the time of randomization. Study interventions may be added or removed according to adaptive design and/or emerging evidence. When there are multiple study interventions available, randomization will occur based on appropriateness of each intervention for the participant as determined by the study protocol.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age at the time of enrollment
2. Previous suspected, probably or confirmed SARS-CoV-2 infection, as defined by the Pan American Health Organization*

   *Suspected and probable cases will only be allowed if it occurred before May 1, 2021, and will be limited to 10% of the study population. Otherwise, confirmed cases are required.

   Suspected case of SARS-CoV-2 infection - Three options, A through C:

   A. A person who meets the clinical OR epidemiological criteria. Clinical criteria: Acute onset of fever AND cough (influenza-like illness) OR Acute onset of ANY THREE OR MORE of the following signs or symptoms: fever, cough, general, weakness/fatigue, headache, myalgia, sore throat, coryza, dyspnea, nausea, diarrhea, anorexia. Epidemiological criteria: Contact of a probable or confirmed case or linked to a COVID-19 cluster; or

   B. Acute respiratory infection with history of fever or measured fever of ≥ 38°C; and cough; with onset within the last 10 days; and who requires hospitalization); or

   C. With no clinical signs or symptoms, NOR meeting epidemiologic criteria with a positive professional use or self-test SARS-CoV-2 antigen-Rapid Diagnostic Test.

   Probable case of SARS-CoV-2 infection:

   A. A patient who meets clinical criteria above AND is a contact of a probable or confirmed case or is linked to a COVID-19 cluster.

   Confirmed case of SARS-CoV-2 infection - Two options, A through B:

   A. A person with a positive nucleic acid amplification test, regardless of clinical criteria OR epidemiological criteria; or

   B. Meeting clinical criteria AND/OR epidemiological criteria (See suspect case A). With a positive professional use or self-test SARS-CoV-2 Antigen-Rapid Diagnostic Test.
3. At least two moderate symptoms from the same symptom cluster or one severe cluster-associated symptom identified via the Cluster Targeted COVID-19 Symptom Questions (CTCSQ), with participant identifying new symptoms since COVID-19 illness and having persisted for at least 12 weeks
4. Meeting PRO Symptom Cluster criteria for at least one Symptom Cluster
5. Willing and able to provide informed consent, complete the surveys, clinical assessments, and return for all of the necessary follow-up visits

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study. Refer to appendices for additional appendix-level criteria:

1. Known active acute SARS-CoV-2 infection ≤ 4 weeks from consent
2. Known severe anemia, defined as < 8 g/dL
3. Meeting the following symptom cluster exclusion for all eligible clusters*:

   a. Cognitive dysfunction: known stroke that resulted in cognitive impairment within 3 months of enrollment b. Autonomic dysfunction: atrial fibrillation or significant cardiac arrhythmia, more than moderate alcohol consumption**, pre-existing sustained severe hypertension (BP> 180/110 mmHg in the sitting position) c. Exercise intolerance: i. any of the following within 4 weeks of consent - an acute myocardial infarction or unstable angina, uncontrolled arrhythmias causing symptoms or hemodynamic compromise, acute myocarditis or pericarditis, uncontrolled acutely decompensated heart failure (acute pulmonary edema), acute pulmonary embolism, suspected dissecting aneurysm, severe hypoxemia at rest, any acute or chronic disorder that may affect exercise performance ii. if the participant is aggravated by exercise (e.g., infection, thyrotoxicosis, unable to cooperate)

   *Participants who are eligible for > 1 cluster must meet all inclusion and no exclusion criteria for an individual symptom cluster. If not, the participant will be excluded from that individual symptom cluster.

   ** Defined as greater than 2 drinks a day for men and 1 drink a day for women. A drink is equivalent to 12 ounces of beer (5% alcohol content), 8 ounces of malt liquor (7% alcohol content), 5 ounces of wine (12% alcohol content), 1.5 ounces or a "shot" of 80-proof (40% alcohol content) distilled spirits or liquor (e.g., gin, rum, vodka, whiskey). 21
4. Known diagnosis of chronic Lyme disease with persistent symptoms, sequelae, or related therapy
5. Any non-marijuana illicit drug use within 30 days of informed consent
6. Current or recent use (within the last 14 days) of study intervention*
7. Known allergy/sensitivity or any hypersensitivity to components of the study intervention (s) or control*
8. Known contraindication(s) to study intervention(s),
9. Inability to discontinue symptomatic medications for the identified time periods
10. Moderate or severe immunocompromised patients, such as those described in the NIH COVID-19 Treatment Guidelines (https://www.covid19treatmentguidelines.nih.gov/ special populations/immunocompromised/)
11. Currently enrolled in another clinical trial outside this platform protocol or another study intervention appendix in this platform protocol***

    ***Participants may re-enroll in the trial for a different study intervention appendix if the participant has completed an appropriate washout period and efficacy has been determined for the appendix in which the participant was previously enrolled.
12. Any condition that would make the participant, in the opinion of the investigator, unsuitable for the study

    * If only one study intervention appendix is open at the time of enrollment. If multiple study intervention appendices are open, a participant may be excluded from any study intervention appendix based on contraindications listed in the study intervention appendix, current use of study intervention, or known allergy/sensitivity/hypersensitivity and still remain eligible for the remaining study intervention appendices.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 963 (Actual)
Dates: Start 2023-07-26 (Actual); Primary Completion 2024-08-06 (Actual); Study Completion 2025-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kanecia Zimmerman, MD PhD, Study Chair — Duke University; Richard Whitley, MD, Study Chair — University of Alabama at Birmingham Medical Center
Locations (69):
- United States (68):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Arizona/Banner University Medical Center Phoenix, Phoenix, Arizona
  - University of Arizona Banner Medical Center, Tucson, Arizona
  - Cedars Sinai Medical Center, Los Angeles, California
  - Hoag Memorial Hospital, Newport Beach, California
  - University of California San Francisco General Hospital, San Francisco, California
  - Stanford University, Stanford, California
  - Los Angeles Biomedical Institute at Harbor-UCLA Medical Center, Torrance, California
  - University of Colorado, Aurora, Colorado
  - Howard University Hospital, Washington D.C., District of Columbia
  - University of Florida College of Medicine Jacksonville, Jacksonville, Florida
  - Lakeland Regional Medical Center, Lakeland, Florida
  - Valencia Medical and Research Center, Miami, Florida
  - Grady Memorial Hospital, Atlanta, Georgia
  - Kaiser Permanente Southwood, Atlanta, Georgia
  - Morehouse School of Medicine, Atlanta, Georgia
  - Atlanta VA Medical Center, Atlanta, Georgia
  - Emory Health Care, Decatur, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - North Shore University Health System, Evanston, Illinois
  - Koch Family Medicine, Morton, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Saint Francis Medical Center, Peoria, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Jadestone Clinical Research, LLC, Silver Spring, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Brigham and Womens Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Washington University School of Medicine, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Rutgers University-Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - University of New Mexico Health Science Center, Albuquerque, New Mexico
  - NYU Langone Health/Brooklyn Hospital, Brooklyn, New York
  - St. Lawrence Health Medical Campus, Canton, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Weil Cornell Medicine, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Duke Clinical and Translational Science Institute, Kannapolis, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Lillestol Research, LLC, Fargo, North Dakota
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - MetroHealth System, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Oklahoma Clinical and Translational Science Institute, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - UPMC Presbyterian Shadyside, Pittsburgh, Pennsylvania
  - Avera McKennan Hospital & University Health Center, Sioux Falls, South Dakota
  - Clinical Trials Center of Middle Tennessee, Franklin, Tennessee
  - Houston Methodist Hospital, Houston, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Vermont Lung Center, University of Vermont, Colchester, Vermont
  - University of Virginia, Charlottesville, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Swedish Health Services, Seattle, Washington
  - University of Washington, Seattle, Washington
  - Providence Medical Research Center, Spokane, Washington
  - West Virginia Clinical and Translational Science Institute, Morgantown, West Virginia
  - Froedtert Hospital-Medical College of Wisconsin, Milwaukee, Wisconsin
- Hispanic Alliance for Clinical and Translational Research, Univ of Puerto Rico, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No
The PIs will share the summary of results on the study website: https://recovercovid.org/

REFERENCES:
- See also: Related Info — http://recovercovid.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a platform study record. Study recruitment period was from late July 2023 to mid-August 2024 at 69 US sites. Recruiting centers were a mix of large academic and small independent research sites in rural and urban, outpatient settings.
Pre-assignment Details: Consented participants were required to endorse two moderate or one severe symptom in one of 3 symptom clusters (exercise intolerance, autonomic dysfunction, or cognitive dysfunction), then meet or exceed a minimal score on a symptom specific questionnaire prior to being assigned. In addition to platform protocol inclusion and exclusion, participants had to meet no symptom cluster exclusion criteria and meet all drug appendix inclusion criteria and no drug appendix exclusion criteria.
Period: Overall Study
Arm/Group | Experimental: Paxlovid 25 Day Dosing | Experimental: Paxlovid 15 Day Dosing | Placebo Comparator: Control
Started | 323 | 320 | 320
Completed | 304 | 297 | 304
Not Completed | 19 | 23 | 16
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Lost to Follow-up | 11 | 10 | 10
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Withdrawal by Subject | 5 | 7 | 6
Not completed — Did Not Meet Eligibility Criteria | 0 | 4 | 0
Not completed — Study Drug Non-compliance | 0 | 1 | 0
Not completed — Moved Out of State Unexpectedly | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Modified Intent to Treat population consists of all randomized participants who receive at least part of one dose of the study intervention or control and who are eligible, enrolled and randomized into a symptom cluster. Prior to protocol version 3, a participant could be randomized into multiple symptom clusters. Therefore, the number of individual participants randomized and the number of slots in a symptom cluster will not match.
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: Paxlovid 25 Day Dosing | Experimental: Paxlovid 15 Day Dosing | Placebo Comparator: Control | Total
Number analyzed (Participants) | 321 | 312 | 318 | 951
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.5 (13.77) | 48.8 (13.89) | 47.1 (14.31) | 48.4 (14.01)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex/Gender: Female | 217 | 209 | 212 | 638
  Sex/Gender: Male | 103 | 102 | 106 | 311
  Sex/Gender: Undifferentiated | 1 | 0 | 0 | 1
  Sex/Gender: Unknown | 0 | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31 | 33 | 44 | 108
  Not Hispanic or Latino | 288 | 277 | 272 | 837
  Unknown or Not Reported | 2 | 2 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 2
  Asian | 19 | 9 | 13 | 41
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 41 | 31 | 37 | 109
  White | 244 | 254 | 249 | 747
  More than one race | 9 | 9 | 8 | 26
  Unknown or Not Reported | 6 | 9 | 10 | 25
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 321 | 312 | 318 | 951

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Participants Enrolled in Each Appendix
Description: Appendix-specific outcome measure data will be reported under the associated NCT ID.
Time Frame: 90 days
Population: Enrolled participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Paxlovid 25 Day Dosing | Experimental: Paxlovid 15 Day Dosing | Placebo Comparator: Control
Number analyzed (Participants) | 323 | 320 | 320
Participants | 323 | 320 | 320

ADVERSE EVENTS:
Time Frame: Up to approximately 90 days
Description: All-cause mortality events and SAEs (Serious Adverse Events) were collected during screening and from start of intervention to end of intervention. Non-serious AEs were not collected during the screening period.
Arm/Group | Experimental: Paxlovid 25 Day Dosing | Experimental: Paxlovid 15 Day Dosing | Placebo Comparator: Control
All-Cause Mortality (participants affected / at risk) | 0/321 | 0/312 | 0/318
Serious Adverse Events (participants affected / at risk) | 0/321 | 0/312 | 0/318
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-18): https://cdn.clinicaltrials.gov/large-docs/69/NCT05595369/Prot_SAP_001.pdf
  • Informed Consent Form (2024-05-30): https://cdn.clinicaltrials.gov/large-docs/69/NCT05595369/ICF_000.pdf